CLINICAL TRIAL: NCT04437680
Title: Retrospective Chart Review Study of Patients Treated With Votiva Device
Status: Completed | Type: Observational
Sponsor: InMode MD Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: DO609635A
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Vulvovaginal Signs and Symptoms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Votiva device — A retrospective chart review of the medical records

SUMMARY:
retrospective data collection is to gain insight into patients satisfaction post Votiva treatments for the complex of vulvovaginal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18years of age at the time of the procedure
* patients with symptoms of at least one of the following: vaginal relaxation syndrome, vaginal atrophy, vaginal dryness, dyspareunia, SUI, Vaginal laxity, recurrent UTI, recurrent vaginal infections, Linchen Sclerosis, perineal pain, itchiness.
* At least one Votiva procedure that included FormaV applicator treatment with or without combination with Fractora/Morpheus8 Applicators treatments

Exclusion Criteria:

* active infection, collagen disorders, immunocompromised state, medications that mitigate inflammatory response, and propensity for keloid/hypertrophic scarring.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — patients with symptoms of at least one of the following: vaginal relaxation syndrome, vaginal atrophy, vaginal dryness, dyspareunia, SUI, Vaginal laxity, recurrent UTI, recurrent vaginal infections, Linchen Sclerosis, perineal pain, itchiness
Study Population: A retrospective chart review of the medical records of 2 practices will be performed by investigators listed in the approved IRB protocol. Patients are seen at 1 site from August 2018 - May 2020, at 2nd site from September 2018 - February 2020 will be included. Patents who have received RF treatment with Votiva will be identified and selected.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Participant satisfaction post treatment | 4 weeks post treatment
  • Participant satisfaction post treatment. Number of patients who are satisfied with post treatment results [ Time Frame: Baseline to 4 weeks post-treatment/s]

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Advanced Women's Care of the Lowcountry, Hilton Head Island, South Carolina
  - Owen Health Group, Lubbock, Texas

IPD SHARING:
Plan to Share IPD: No